CLINICAL TRIAL: NCT00291798
Title: Neoadjuvant Endocrinotherapy of Mamma Carcinoma With Exemestane
Brief Title: Neoadjuvant Endocrinotherapy of Breast Cancer (Mamma Carcinoma) With Exemestane
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Pharmacia Austria GmbH (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG-17
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-02

CONDITIONS: Breast Cancer
Keywords: pilot study; exemestane; endocrinotherapy; mamma carcinoma; neoadjuvant; ABCSG; 17
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: rate of remission

SUMMARY:
The objective of the present clinical investigation is to determine whether hormonal therapy given preoperatively is able to reduce tumor size to an extent that facilitates breast-conserving procedures.

DETAILED DESCRIPTION:
This open, prospective multicenter Phase II pilot trial investigates the efficacy of exemestane, 25 mg once daily over 4 months, in postmenopausal women with primary breast cancer, measured in terms of clinical response

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified breast cancer (punch biopsy), established HER-2/neu status
* Postmenopausal patients (> 1 year following outset of menopause and/or postmenopausal hormonal profile)
* Clinical staging: T2 (> 3 cm), T3, T4a-c, N0-1
* Hormone receptor positivity, i.e. estrogen and/or progesterone receptor > 10 fmol/mg cytosolic protein or ER-ICA-positive and/or PgR-ICA-positive. Positivity of + (low-grade) in one hormone receptor is only eligible in the presence of positivity in the other hormone receptor.
* no internal contraindication
* life expectation > 6 month
* written informed consent

Exclusion Criteria:

* premenopausal patients and patients with no clearly indicated menopausal status
* manifest second malignant tumor (except basalioma or in situ carcinoma of cervix uteri)
* uncontrolled internal disease i.e. diabetes mellitus, cardiac disease (NYHA III/IV)
* thromboembolic disease
* inflammatory mamma carcinoma
* existence of distant metastases
* former or simultaneously therapy with antioestrogens, aromatase inhibitors, cytostatics or radiotherapy
* corticosteroids before and during the study (except inhalant application)
* lack of compliance

Min Age: 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98
Dates: Start 2000-09; Study Completion 2009-03

PRIMARY OUTCOMES:
rate of remission

SECONDARY OUTCOMES:
Toxicity (WHO-grading)
rate of mastectomy
response of tumor subject to HER2-status
collection of disease free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Mlineritsch, MD, Study Chair — Austrian Breast & Colorectal Cancer Study Group
Locations (11):
- Austria (11):
  - Hospital of Guessing, Güssing, Burgenland
  - State Hospital Klagenfurt, Surgery, Klagenfurt, Carinthia
  - State Hospital Wolfsberg, Wolfsberg, Carinthia
  - Hospital of Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Paracelsus Medical University Salzburg, Oncology, Salzburg, Salzburg
  - Gynaegological Medical University of Graz, Graz, Styria
  - Medical University of Graz, Oncology, Graz, Styria
  - Hospital BHS Linz, Linz, Upper Austria
  - General Hospital Linz, Linz, Upper Austria
  - Medical University of Vienna, General Hospital, Vienna, Vienna
  - Hanusch Hospital, Vienna, Vienna

REFERENCES:
- See also: Related Info — http://www.abcsg.at